CLINICAL TRIAL: NCT04822766
Title: Allogeneic Hematopoietic Cell Transplantation Versus Best Available Standard of Care Therapy in Elderly Patients With Acute Myeloid Leukemia: a Randomized Phase 3 Trial
Brief Title: A Study Comparing Allogeneic Hematopoietic Cell Transplantation Versus Best Available Standard of Care Therapy in Elderly Patients With Acute Myeloid Leukemia
Acronym: ALLO-BEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200134; 2020-A01456-33 (Other: ANSM)
Record Dates: First submitted 2021-01-24; First posted 2021-03-30 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Allogeneic; hematopoietic cell transplantation; acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy (Active Comparator)
  Interventions: Drug: Best chemotherapy treatment
- Allogeneic Hematopoietic Cell Transplantation (Experimental): Time of transplant procedure The best available treatments of AML
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — patients will undergo allo-HSCT after consolidation therapy (or completion of other appropriate non-palliative strategy) according to standard procedures of the transplant center (choice of donor, conditioning regimen, GVHD and infection prophylaxis). The use of novel therapies (such as sorafenib, midaustorine, venetoclax, etc.) will be allowed as post-transplantation maintenance strategy.
  Arms: Allogeneic Hematopoietic Cell Transplantation
Drug: Best chemotherapy treatment — patients will be treated according to the standard procedures of the treating center for this type of population. Patients will receive the best available treatments (including additional conventional chemotherapy or other non-palliative therapies such as 5-azacytidine, decitabine, venetoclax, midaustorine, enasidenib, etc.).
  Arms: Chemotherapy

SUMMARY:
A subject of major interest for researchers, clinicians, patients, and payers, is the role of allogeneic hematopoietic stem cell transplantation (allo-HSCT) in the treatment of these older patients with AML. With conventional induction chemotherapy or hypomethylating agents, the expected 2-year overall survival (OS) is less than 25% in patients with intermediate- or high-risk disease. The 2-year OS ranges from 50 to 56% with allo-HSCT in AML patients older than 65 years.

Performing an allo-HSCT in older patients is however still controversial because of the higher risk of non-relapse mortality (15 to 35%) and graft-versus-host disease. Depending on the center policy, patients older than 65 years will either be contraindicated for transplant or will receive allo-HSCT.

With a phase III comparative, randomized, controlled, prospective, multicenter study, the trial aim to assess prospectively the outcomes and quality of life of older patients with AML receiving allo-HSCT strategy compared to those receiving a non-transplant approach.

DETAILED DESCRIPTION:
Every year, 30,000 patients in Europe and 20,000 in the USA are diagnosed with acute myeloid leukemia (AML). More than half of them are over 65 years old. In this older population, the median overall survival (OS) is only 2 to 8 months. With conventional induction chemotherapy or hypomethylating agents, the expected 2-year OS is less than 25% in patients with intermediate- or high-risk disease.

Performing an allo-HSCT in older patients is however still controversial because of the higher risk of non-relapse mortality (15 to 35%) and graft-versus-host disease. Depending on the center policy, patients older than 65 years will either be contraindicated for transplant or will receive allo-HSCT. Noteworthy, no prospective randomized trial has yet compared allo-HSCT to a non-transplant strategy in older patients with AML. A previous attempt made 10 years ago, by the EBMT to run a slightly similar trial, has failed in France and most European countries, mainly (i) because it mandated the type of transplant procedure to be applied and (ii) because of the absence of novel and effective drugs.

Every year, 30,000 patients in Europe and 20,000 in the USA are diagnosed with acute myeloid leukemia (AML). More than half of them are over 65 years old. In this older population, the median overall survival (OS) is only 2 to 8 months. With conventional induction chemotherapy or hypometylating agents, the expected 2-year OS is less than 25% in patients with intermediate- or high-risk disease.

Performing an allo-HSCT in older patients is however still controversial because of the higher risk of non-relapse mortality (15 to 35%) and graft-versus-host disease. Depending on the center policy, patients older than 65 years will either be contraindicated for transplant or will receive allo-HSCT. Noteworthy, no prospective randomized trial has yet compared allo-HSCT to a non-transplant strategy in older patients with AML. A previous attempt made 10 years ago, by the EBMT to run a slightly similar trial, has failed in France and most European countries, mainly (i) because it mandated the type of transplant procedure to be applied and (ii) because of the absence of novel and effective drugs.

New targeted therapies and treatment strategies are evolving rapidly. A standardized unique treatment administrated to all sub-types of AML is no longer the optimal approach for induction and non-transplant maintenance strategies. No treatment has reached consensus for older patients. For these reasons, this trial will not limit the choices of drugs administered to the patients but compare two strategies allowing patients to receive the best available standard of care.

The trial aim to assess prospectively the outcomes and quality of life of older patients with AML receiving allo-HSCT strategy compared to those receiving a non-transplant approach.

Patients will receive initial treatment with chemotherapy (or other appropriate non-palliative therapy). Once first complete remission is achieved and a donor is identified, patients will be included.

Patients will be randomly assigned (1:1) after inclusion to receive one of the following strategy:

* Allogeneic hematopoietic stem cell transplantation arm: patients will undergo allo-HSCT after consolidation therapy (or completion of other appropriate non-palliative strategy) according to standard procedures of the transplant center (choice of donor, conditioning regimen, GVHD and infection prophylaxis). The use of novel therapies (such as sorafenib, midaustorine, venetoclax, etc.) will be allowed as post-transplantation maintenance strategy
* Non-transplant arm: patients will be treated according to the standard procedures of the treating center for this type of population.

All patients will receive the best available treatments (including additional conventional chemotherapy or other non-palliative therapies such as 5-azacytidine, decitabine, venetoclax, midaustorine, enasidenib, etc.). Supportive care will be performed according to each participating center usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age ≥ 65 and ≤ 75 years
* Newly diagnosed patients with de novo or secondary AML in first complete remission who are considered as potential candidates and eligible for an allo-HSCT procedure
* Presence of a donor (matched related or unrelated or haplo-mismatched) willing to donate peripheral blood stem cells
* Patient is fit for the allo-HSCT procedure
* Patient is fit for further consolidation therapy (non-transplant arm)
* Written informed consent

Exclusion Criteria:

* Acute promyelocytic leukemia (AML FAB M3)
* AML deemed not eligible for allo-HSCT
* Karnofsky score <70%
* HIV positive patient
* Life expectancy less than one month according to the attending physician
* Acute or chronic heart failure (Cardiac ejection fraction < 40%)
* Pulmonary function - diffusion capacity < 50% predicted
* Estimated glomerular filtration rate < 50 ml/min (CKD-EPI)
* Severe neurological disorders
* Patient subject to a legal protection measure (guardianship, curatorship and safeguard of justice) or unable to consent
* Patient deprived of their liberty by a judicial or administrative decision
* Patient with severe psychiatric disorders or hospitalized without consent for psychiatric care

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years after the inclusion
  From inclusion (time of identification of potential donor) until death or at 24 months, whichever comes first]

SECONDARY OUTCOMES:
Leukemia free survival | within the 2 years after inclusion
  from inclusion (time of identification of potential donor) until relapse and/or death from any cause or at 24 months, whichever comes first
Assessment of MRD and time to relapse from inclusion up to 2 years | : time between inclusion and date of relapse or at 24 months, whichever comes first]
Quality of life FACT-BMT | at baseline, 12 and 24 months after inclusion
  FACT-BMT (Functional Assessment of Cancer Therapy - Bone Marrow Transplant)
Quality of life EQ 5D 5L | at baseline, 12 and 24 months after inclusion
  EQ 5D 5L (EuroQol group)
The Incremental cost-effectiveness ratios (ICERs) expressed in cost per quality-adjusted life-year (QALY) gained | 2 years after inclusion
  from inclusion (time of identification of potential donor) until death from any cause or at 24 months, whichever comes first
The Incremental cost-effectiveness ratios (ICERs) expressed in cost per Life Year Gained | 2 years after inclusion
  from inclusion (time of identification of potential donor) until death from any cause or at 24 months, whichever comes first
Non-relapse mortality | within the 2 years after inclusion
  from inclusion (time of identification of potential donor) until death without evidence of relapse or at 24 months, whichever comes first
In allo-HSCT patients only: cumulative incidence of acute and chronic graft-versus-host disease (GVHD) | within the 2 years after inclusion
  from transplantation until occurrence of GVHD or death from any cause or at 24 months after inclusion, whichever comes first
In allo-HSCT patients only: severity of acute and chronic graft-versus-host disease (GVHD) | within the 2 years after inclusion
  from transplantation until occurrence of GVHD or death from any cause or at 24 months after inclusion, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Rémy DULERY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital - Hematology Department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided